CLINICAL TRIAL: NCT00558311
Title: A Prospective, Multi-center, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Assess the Efficacy and Safety of Clazosentan in Reducing Vasospasm-related Morbidity and All-cause Mortality in Adult Patients With Aneurysmal Subarachnoid Hemorrhage Treated by Surgical Clipping.
Brief Title: Clazosentan in Reducing Vasospasm-related Morbidity and All-cause Mortality in Adult Patients With Aneurysmal Subarachnoid Hemorrhage Treated by Surgical Clipping
Acronym: CONSCIOUS-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-054-301
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
Keywords: Aneurysmal; Subarachnoid; Hemorrhage; vasospasm; clazosentan; PIVLAZ; surgical clipping
MeSH Terms: conditions — Subarachnoid Hemorrhage; Hemorrhage | interventions — clazosentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clazosentan (Experimental): A continuous intravenous infusion of clazosentan was started within 56 hours post-aSAH and was scheduled to continue during the hospitalization until Day 14 post-aSAH, or at least until Day 10.
  Interventions: Drug: Clazosentan
- Placebo (Placebo Comparator): A continuous intravenous infusion of placebo-matching clazosentan was started within 56 hours post-aSAH and was scheduled to continue during the hospitalization until Day 14 post-aSAH, or at least until Day 10.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clazosentan — Intravenous clazosentan administered by continuous infusion at 5 mg/h
  Arms: Clazosentan
Drug: Placebo — Placebo administered by continuous infusion matching clazosentan administration
  Arms: Placebo

SUMMARY:
The aim of this study is to demonstrate that clazosentan, administered as a continuous intravenous infusion at 5 mg/h until Day 14 post aneurysmal subarachnoid hemorrhage (aSAH), reduces the incidence of cerebral vasospasm -related morbidity and all-cause mortality within 6 weeks post-aSAH treated by surgical clipping. The primary endpoint of the study is the occurrence of cerebral vasospasm-related morbidity, and mortality of all-causes within 6 weeks post-aSAH, defined by at least one of the following:

1. Death (all causes).
2. New cerebral infarct(s) due to cerebral vasospasm as either the primary or relevant contributing cause, or not adjudicated to be entirely due to causes other than vasospasm.
3. Delayed ischemic neurological deficit (DIND) due to cerebral vasospasm as either the primary or relevant contributing cause, or not adjudicated to be entirely due to causes other than vasospasm.
4. Neurological signs or symptoms (depending on state of consciousness), in the presence of confirmed cerebral vasospasm on angiography (DSA or CTA), leading to the administration of a valid rescue therapy.

An independent Critical Events Committee (CEC) will adjudicate whether or not patients meet the primary endpoint and its individual morbidity components.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18 to 75 years (inclusive).
2. Patients with a ruptured saccular aneurysm, confirmed by angiography (digital subtraction angiography [DSA] or computed tomography angiography [CTA]), and which has been successfully secured by surgical clipping. The time of aneurysm rupture must be known or possible to estimate with a reasonable degree of certainty.
3. World Federation of Neurological Surgeons (WFNS) grade I-IV measured prior to the clipping procedure, and which does not worsen to grade V post-procedure (based on regular Glasgow Coma Scale [GCS])*
4. Patients with any diffuse clot (long axis > or = 20 mm, or any clot present across both hemispheres) on baseline CT scan.
5. Women of childbearing potential must have a negative serum pregnancy test and must use a reliable method of contraception during the 12 weeks following study drug discontinuation.
6. Written informed consent to participate in the study must be obtained from the patient or a legal representative prior to initiation of any study-mandated procedure and randomization.

   * Patients must be evaluable for WFNS grade prior to the clipping procedure. Patients who cannot be assessed for WFNS post-procedure due to a requirement for uninterrupted sedation (e.g., for high or unstable intracranial pressure [ICP]) may be included in the study provided that a CT scan is performed at 12 hours post-procedure, but prior to randomization, ruling out any large procedure-related infarct.

Exclusion Criteria:

1. Patients with subarachnoid hemorrhage (SAH) due to causes other than a saccular aneurysm (e.g., trauma or rupture of fusiform or mycotic aneurysms).
2. Patients with intraventricular or intracerebral blood, in the absence of subarachnoid blood, or with only a local clot.
3. Presence of cerebral vasospasm seen on angiography prior to the clipping procedure.
4. Patients who experienced a major complication during the clipping procedure, such as massive bleeding, major arterial occlusion, a large territorial cerebral infarct defined as involving > 1/3 of a vascular territory, or a new major neurological deficit post-procedure (e.g., hemiplegia or aphasia lasting > or = 12 hours post-aneurysm clipping).*
5. Patients for whom study drug cannot be started within 56 hours after the aneurysm rupture.
6. Patients who have had their aneurysm secured by coiling only.
7. Patients for whom it is known, at the time of screening, that certain follow-up, protocol-mandated imaging assessments will not be feasible.
8. Patients with hypotension (systolic blood pressure (SBP)< or = 90 mmHg) that is refractory to treatment.
9. Patients with aspiration pneumonia.
10. Patients with pulmonary edema or severe cardiac failure requiring inotropic support.
11. Any severe or unstable concomitant condition or disease (e.g., known significant neurological deficit, cancer, hematological, or coronary disease), or chronic condition (e.g., psychiatric disorder), which, in the opinion of the investigator, would affect the assessment of the safety or efficacy of the study drug.
12. Significant kidney and/or liver disease, as defined by plasma creatinine > or = 2.5 mg/dL (221 micromol/l) and/or total bilirubin > 3 mg/dL (51.3 micromol/l) measured at the local site laboratory.
13. Patients receiving i.v. nimodipine, i.v. nicardipine, or fasudil hydrochloride, must have these drugs discontinued at least 4 hours prior to initiation of the study treatment.
14. Patients receiving statins for less than 2 weeks prior to admission must have them discontinued prior to study drug initiation.
15. Patients receiving cyclosporin A or other calcineurin inhibitors (e.g., tacrolimus), or patients for whom it is known at the time of randomization that these medications will be started during the study drug infusion period.
16. Patients who have received an investigational product within 28 days prior to randomization or those who have already participated in the current study.
17. Patients unlikely to comply with the protocol (e.g., unable to return for follow-up visits).
18. Known hypersensitivity to other endothelin receptor antagonists.
19. Patients with current alcohol or drug abuse or dependence.

    * Further detail on exclusion criterion number 4:

      * "Large territorial infarct" refers to those infarcts detected during the clipping procedure or immediately post-procedure (i.e., CT performed for suspicion of cerebral infarct or other complication). This does not imply having to wait 24-48 hours post-procedure to perform the protocol-mandated CT scan in order to randomize a patient.
      * Evaluation for a new major neurological deficit post-procedure implies the reversal of sedation (or waiting for the patient to recover from sedation) and the performance of a GCS examination (verbal scores in intubated patients may be extrapolated from the eye-opening and motor scores using the values provided in the table included in Section 3.9.1.2.1 of the protocol). In the event of a new major neurological deficit that does not improve within 12 hours after the clipping procedure, the patient cannot be included in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1157 (Actual)
Dates: Start 2007-12-14; Primary Completion 2010-06-15 (Actual); Study Completion 2010-07-13 (Actual)

PRIMARY OUTCOMES:
Cerebral vasospasm-related morbidity and mortality of all-causes as defined by the protocol | Within 6 weeks post-aSAH

SECONDARY OUTCOMES:
Glasgow Outcome Scale Extended (GOSE) at Week 12 post-aSAH, dichotomized into good (score > 4) and poor (score ≤ 4) outcome. | Week 12 post-aSAH

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (117):
- United States (11):
  - Barrow Neurosurgical Associates, Phoenix, Arizona
  - Colorado Neurological Institute, Englewood, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - State University of New York at Stony Brook-Health Sciences Center, Stony Brook, New York
  - University of Cincinnati-Department of Neurosurgery, Cincinnati, Ohio
  - University Hospitals Case Medical Center-Department of Neurosurgery, Cleveland, Ohio
  - Oregon Health & Science University-Oregon Stroke Center, Portland, Oregon
  - Thomas Jefferson University School of Medicine-Jefferson Hospital for Neuroscience, Philadelphia, Pennsylvania
  - University of Virginia Health System-Department of Neurosurgery, Charlottesville, Virginia
  - Virginia Commonwealth University-Department of Neurosurgery, Richmond, Virginia
- Australia (2):
  - Royal Brisbane Hospital, Herston
  - The Alfred Hospital, Melbourne
- Austria (6):
  - Landeskrankenhaus, Feldkirch
  - Landeskrankenhaus und Medizinische Universitat Graz, Graz
  - Medizinsche Universitat, Innsbruck
  - University Fur Neurochirurgie, SALK, Christian Doppler Hospital, Salzburg
  - AKH University of Vienna, Medical University, Vienna
  - Sozialmedizinisches Zentrum Ost (ZMZ-Ost) Donauspital Vienna, Vienna
- Cliniques Universitaires Saint-Luc, Universite Catholique de, Brussels, Belgium
- Canada (7):
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver Hospital, Vancouver, British Columbia
  - St Michael's Hospital, University, Toronto, Ontario
  - CHUM Notre Dame, Montreal, Quebec
  - University of Calgary Foothills Medical Center, Calgary
  - QEII Health Science Center, Halifax
  - Toronto Western Hospital, University of Toronto, Toronto
- China (6):
  - Beijing Tian Tan Hospital, Beijing
  - XuanWu Hospital Institute of Brain Vascular Disease, Beijing
  - Guangdong Province Chinese Medicine Hospital, Guangzhou
  - 1st Affilated Hospital of Zhongshan, Guangzhou
  - Shanghai Hua Shan Hospital, Shanghai
  - Wuhan Tongji Hospital, Wuhan
- Croatia (3):
  - Clinical Hospital "Dubrava", Zagreb
  - Clinical Hospital Dubrava, Zagreb
  - University Hospital Sestre Milosrdnice, Zagreb
- Czechia (4):
  - Faculty Hospital/FN Brno Bohunice, Brno
  - Nemocnice Ceske Budejovice, České Budějovice
  - Na Homolce Hospital Prague, Prague
  - UVN Prague, Prague
- Denmark (3):
  - Copenhagen University Hospital, Copenhagen
  - Copenhagen Country Hospital, Glostrup Municipality
  - Odense University Hospital, Odense
- Finland (3):
  - Helsinki University Central Hospital, Helsinki
  - Oulu University Hospital, Oulu
  - Tampere University Central Hospital, Tampere
- France (5):
  - Pole d'Anesthesie Reanimation, CHU D'Angers, Angers
  - Hopital Pellegrin, Bordeaux
  - Hopital Neurologique et Neuro-Chirurgical Pierre Wertheimer, Bron
  - Chu Hopital Gabriel Montpied, Clermont-Ferrand
  - Hopital de la Timone, Marseille
- Germany (12):
  - Charite Universitatsmedizin Berlin-Neurochirurgische Klinik-CVK, Berlin
  - University of Bonn Medical Center, Bonn
  - Klinik und Poliklinik fur Neurochirurgie, Dresden
  - University of Erlangen-Nurnberg, Erlangen
  - University of Hospital of Essen, Essen
  - Universitatsklinik Frankfurt, Klinik und Poliklinik fur Neurochirurgie, Frankfurt
  - University Hospital of Hamburg, Hamburg
  - Neurochirurggische Universitatsklinik des Heidelberg, Heidelberg
  - Klinik und Poliklinik fur Neurochirurgie, Leipzig
  - University Munich Groshadern, Munich
  - Thechnical University-Klinikum rechts der Isar, Munich
  - University Regensburg, Regensburg
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- India (6):
  - Post Graduate Institute of Medical Education and Research, Chandigarh
  - Post Graduate Institute of Medical Education, Chandigarh
  - Nizam's Institute of Medical Sciences, Hyderabaad
  - All India Insititute of Medicla Sciences (AIIMS), New Delhi
  - Sahyadri Specialty Hospital, Pune
  - Sahyadri Hospital, Pune
- Italy (8):
  - Ospedale Bellaria-Maggiore Hospital, Bologna
  - Ospedale Maurizio Bufalini, Cesena
  - Azienda Ospedaliero-Universitaria di Careggi, Florence
  - Ospedale Niguarda, Milan
  - Nuovo Ospedale Sant' Agostino Estense, Modena
  - Ospedale Civile di Padova, Padua
  - Azienda Ospedaliero-Universitaria di, Parma
  - Ospedale Civile Borgo Trento, Verona
- Riga Eastern Clinical University Hospital, Riga, Latvia
- Auckland Hospital, Grafton, New Zealand
- Norway (3):
  - Haukeland University Hospital Helse Bergen HF, Bergen
  - Ulleval University Hospital, Oslo
  - Universitetssykehuset Nord-Norge, Tromsø
- Poland (8):
  - Klinika Neurochirurgii AMB-Neurosurgery Clinic of Medical Academy, Bialystok
  - Kathedra I Klinika Neurochirurghii I Neurotraumatologii Collegium Medicum im. L. Rydygiera w Bydgoszc, Bydgoszcz
  - Katedra Klinika Neurochirurgii Akademii Medycznej w Gdansku, Gdansk
  - Samodzielny Publiczny Szpital Kliniczny Slaskiej Akademii Medycznej w Katowicach, Katowice
  - Oddzial Kliniczny Kliniki Neurochirurgii i Neurotrumatologii Szpitala, Uniwersyteckiego w Krakowie, Krakow
  - Katedra Neurochirurgii, Uniwersytet, Lodz
  - Katedra I Klinika Neurochirurgii i Dzieciecej, Lublin
  - Katedra IKlinika Neurochirurgii Akademii Medycznej w Warszawie Clinic, Warsaw
- Scientific Research Institute of Neurosurgery by Burdenko, Moscow, Russia
- Serbia (2):
  - Clinical Center Nis, Niš
  - Clinical Center Novi Sad, Novi Sad
- National Neuroscience, Singapore, Singapore
- General Hospital Maribor, Maribor, Slovenia
- South Korea (2):
  - Kyungpook National University, Daegu
  - Daejeon Eulji University Hospital, Daejeon
- Spain (4):
  - Hospital Del Mar, Barcelona
  - Vall d'Hebron Hospital, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital de Son Dureta, Palma de Mallorca
- Sweden (3):
  - Sahlgrenska, Gothenburg
  - Lund University Hospital, Lund
  - Uppsala University Hospital-Uppsala Akademiska Sjukhus, Uppsala
- Switzerland (6):
  - Kantonsspital Aarau, Aarau
  - Universitatsklinik Bern, Bern
  - Universitätsklinik Bern Klinik für Neurochirurgie, Bern
  - Geneva University Hospital, Geneva
  - Kantonsspital St. Gallen, Sankt Gallen
  - Universitatsspital Zurich, Zurich
- Turkey (Türkiye) (3):
  - Ibn-i Sina Hastanesi Ankara & Ankara Universitesi Tip Fakultesi, Ankara
  - Ege Universitesi Tip Fak Hestanesi, Bornova
  - Istanbul Universitesi, Istanbul Tip, Istanbul
- Ukraine (2):
  - Regional Clinical Hospital by Mechnikov, Dnipropetrovsk
  - A. P. Romodanov Institute of Neurosurgery, Kiev

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mayer SA, Aldrich EF, Bruder N, Hmissi A, Macdonald RL, Viarasilpa T, Marr A, Roux S, Higashida RT. Thick and Diffuse Subarachnoid Blood as a Treatment Effect Modifier of Clazosentan After Subarachnoid Hemorrhage. Stroke. 2019 Oct;50(10):2738-2744. doi: 10.1161/STROKEAHA.119.025682. Epub 2019 Aug 9. PMID 31394993
- [Derived] Macdonald RL, Higashida RT, Keller E, Mayer SA, Molyneux A, Raabe A, Vajkoczy P, Wanke I, Bach D, Frey A, Marr A, Roux S, Kassell N. Randomised trial of clazosentan, an endothelin receptor antagonist, in patients with aneurysmal subarachnoid hemorrhage undergoing surgical clipping (CONSCIOUS-2). Acta Neurochir Suppl. 2013;115:27-31. doi: 10.1007/978-3-7091-1192-5_7. PMID 22890639
- [Derived] Macdonald RL, Higashida RT, Keller E, Mayer SA, Molyneux A, Raabe A, Vajkoczy P, Wanke I, Bach D, Frey A, Marr A, Roux S, Kassell N. Clazosentan, an endothelin receptor antagonist, in patients with aneurysmal subarachnoid haemorrhage undergoing surgical clipping: a randomised, double-blind, placebo-controlled phase 3 trial (CONSCIOUS-2). Lancet Neurol. 2011 Jul;10(7):618-25. doi: 10.1016/S1474-4422(11)70108-9. Epub 2011 Jun 2. PMID 21640651